CLINICAL TRIAL: NCT01578772
Title: Telmisartan and Flow-Mediated Dilatation in Older HIV-Infected Patients at Risk for Cardiovascular Disease
Brief Title: A Clinical Trial for People HIV+ Age > 50 at Risk for Heart Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: The Campbell Foundation (Other)
Responsible Party: Principal Investigator, Jordan E. Lake M.D., M.D., University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: miFMD
Record Dates: First submitted 2012-02-01; First posted 2012-04-17 (Estimated); Results first posted 2014-12-08 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Endothelial Dysfunction
Keywords: HIV; Flow-mediated dialation (FMD); Telmisartan; Cardiovascular disease (CVD); HIV+ men and women age > 50 at risk for heart disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Telmisartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Telmisartan (Experimental): Open label
  Interventions: Drug: Telmisartan

INTERVENTIONS:
Drug: Telmisartan — 80mg tablets po daily for 6 weeks
  Other Names: Micardis

SUMMARY:
This research study is to see whether blood vessel function, an early sign of heart disease, improves in HIV-infected men and women who take telmisartan for 12 weeks. The investigators will be looking at how a blood vessel in the arm, called the brachial artery, changes in response to stress before and after taking telmisartan. To determine how well the blood vessel functions, the investigators will be using an ultrasound machine.

Telmisartan is not an HIV medication. It is an FDA-approved medication designed to treat blood pressure, but has been shown to improve blood vessel function in HIV-negative people with and without high blood pressure. Telmisartan is made by Boehringer Ingelheim, and this trial is sponsored by The Campbell Foundation.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive men and women > 50 years of age.
* HIV-1 RNA documented to be < 50 copies/mL at screening and undetectable by assay of choice (< 50 or < 400 copies/mL) for at least 12 weeks prior to entry.
* Current ART with a suppressive, highly active regimen. Subjects must not have changed ART in the 12 weeks prior to entry, and must not be planning to change ART for the 12-week study duration.
* Systolic blood pressure > 110mmHg.
* One or more risk factors for CVD (smoking, hypertension, hyperlipidemia, diabetes mellitus). Note: family history of early heart disease alone will not be a sufficient entry criterion.
* Ability and willingness of subject to provide informed consent.

Exclusion Criteria:

* Pregnancy (current or within the past 6 months) or nursing.
* Uncontrolled hypertension:
* Prohibited concomitant medications: Other members of the angiotensin receptor-blocking class (losartan, irbesartan, olmesartan, valsartan, candesartan; wash-out period allowed), nelfinavir, and etravirine. Subjects taking nelfinavir or etravirine will be excluded due to the possibility of increased drug levels via inhibition of cytochrome P-450 2C19.

Note 1: Subjects requiring amifostine or rituximab must be aware of the increased risk of orthostatic hypotension with the addition of telmisartan. Any subject requiring lithium therapy while on study must have lithium levels monitored closely by their outside physician. All subjects on the above listed medications should provide documentation that their physician is aware of the study protocol.

Note 2: Subjects taking thiazolidinediones must be on stable dosing (> 12 weeks) and must agree to refrain from dose titration for the 12-week study duration.

* Untreated hyperlipidemia: Subjects must be willing to abstain from initiating therapy for the 12-week study duration. Subjects on a stable (> 12 weeks) lipid-lowering regimen must be willing to remain on their current dose for the 12-week study duration.
* Subjects undergoing treatment for diabetes with oral hypoglycemic agents must be willing to remain on their current dose of insulin-sensitizing agents (metformin/biguanides) for the 12-week study duration. Titration of other diabetes (except thiazolidinediones, see 4.2.3) medications will be permitted.
* Screening laboratory values as follows:
* ANC < 750 cells/mm3
* Hemoglobin < 10 gm/dL
* Creatinine clearance < 30 mL/min (estimated by Cockcroft-Gault equation using ideal body weight)
* AST or ALT > 3 times ULN
* Known, untreated, renal artery stenosis.
* Unstable coronary artery disease/angina, decompensated congestive heart failure, or predicted need for cardiovascular surgery within the study period.
* History of intolerance to any member of the angiotensin receptor blocker class of agents.
* Need for ongoing potassium supplementation.
* Active, untreated opportunistic and/or AIDS-defining illnesses.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan E. Lake, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA CARE Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Lake JE, Seang S, Kelesidis T, Currier JS, Yang OO. Telmisartan increases vascular reparative capacity in older HIV-infected adults: a pilot study. HIV Clin Trials. 2016 Nov;17(6):225-232. doi: 10.1080/15284336.2016.1234222. Epub 2016 Sep 23. PMID 27658740

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Telmisartan
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: HIV-infected individual >50 years old with HIV-1 RNA <50 copies /mL on stable ART and >=1 CVD risk factor.
Arm/Group | Telmisartan
Number analyzed (Participants) | 17
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60 [54 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 15

OUTCOME MEASURES:

1. Primary Outcome: 6-week Change in Diameter and Flow Mediated Dilatation (FMD) of the Brachial Artery With Telmisartan Therapy
Description: Flow-mediated dilatation (FMD) testing of the brachial artery was performed for all participants on Telmisartan treatment at baseline and 6 weeks.
Time Frame: 6 weeks (after baseline)
Measure: Median (Inter-Quartile Range); unit: mm
Groups:
- Baseline (Week 0); Week 6: All participants received telmisartan 80mg tablets po daily for 6 weeks. Flow-mediated dilatation (FMD) testing was performed for all participants at baseline (week 0) and 6 weeks.
Arm/Group | Baseline (Week 0) | Week 6
Number analyzed (Participants) | 17 | 17
mm
  Brachial Artery Diameter | 4.6 [4.4 to 4.9] | 4.7 [4.4 to 5.1]
  Maximum Absolute FMD | 0.1 [0.1 to 0.2] | 0.2 [0.1 to 0.3]
Statistical Analysis 1: Comparison: Baseline (Week 0) vs Week 6; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney); Pairwise comparisons were performed using Wilcoxon signed rank test. All statistical tests are two-sided with nominal alpha level of 0.05; Median Difference (Net) = 0, 95% CI 2-sided [-0.1 to 0.1]

2. Primary Outcome: 6-week Change in Maximum Relative Flow Mediated Dilatation (FMD) of the Brachial Artery With Telmisartan Therapy
Description: as for outcome 1
Time Frame: 6 weeks (after baseline)
Measure: Median (Inter-Quartile Range); unit: percentage of maximum relative FMD
Arm/Group | Baseline (Week 0) | Week 6
Number analyzed (Participants) | 17 | 17
percentage of maximum relative FMD | 2.7 [1.4 to 3.9] | 3.5 [1.6 to 6.0]
Statistical Analysis 1: Comparison: Baseline (Week 0) vs Week 6; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney); [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = 0.7, 95% CI 2-sided [-1.3 to 1.9]

ADVERSE EVENTS:
Time Frame: 6 weeks (after baseline)
Arm/Group | Telmisartan
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

LIMITATIONS AND CAVEATS:
Given the limited size of the study population, the study was underpowered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No